CLINICAL TRIAL: NCT01569126
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY110140 in Healthy Japanese Male Subjects
Brief Title: A Study of LY110140 in Healthy Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14638; B1Y-JE-HCLX (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 5 milligrams (mg) LY110140 (SD) (Experimental): 5 mg administered once in the fasted state on Day 1
  Interventions: Drug: LY110140
- 20 mg LY110140 (SD) (Experimental): 20 mg administered once in the fasted state on Day 1
  Interventions: Drug: LY110140
- 40 mg LY110140 (SD) (Experimental): 40 mg administered once in the fasted state on Day 1
  Interventions: Drug: LY110140
- Placebo (MD) (Placebo Comparator): Placebo once daily oral dosing for 28 consecutive days
  Interventions: Drug: Placebo
- 20 mg LY110140 (MD) (Experimental): 20 mg once daily oral dosing for 28 consecutive days
  Interventions: Drug: LY110140
- 40 mg LY110140 (MD) (Experimental): 40 mg once daily oral dosing for 28 consecutive days
  Interventions: Drug: LY110140

INTERVENTIONS:
Drug: LY110140 — Administered orally as capsules
  Other Names: Fluoxetine Hydrochloride, Prozac, Sarafem
  Arms: 20 mg LY110140 (MD); 20 mg LY110140 (SD); 40 mg LY110140 (MD); 40 mg LY110140 (SD); 5 milligrams (mg) LY110140 (SD)
Drug: Placebo — Administered orally as capsules in the placebo arm and to maintain the blind in the 20 mg LY110140 (MD) arm
  Arms: Placebo (MD)

SUMMARY:
The purposes of this study are to look at safety, how well the study drug (LY110140) is tolerated, and how much of the study drug gets into the blood stream when given as single dose (SD) and multiple doses (MD) to healthy Japanese male participants. Participants will participate in SD portion for approximately 6 weeks and in MD portion for approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy Japanese males (as determined by medical history and physical examination) who agree to use a reliable method of birth control during the study and for 3 months following the last dose of the investigational product.
* Have a body mass index (BMI) of 18.5 to 29.9 kilograms per square meter (kg/m^2), inclusive, at the time of screening.
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the study site.

Exclusion Criteria:

* Poor metabolizers of isoenzyme cytochrome P450 2D6 (CYP2D6) (assessed at screening).
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening that, in the opinion of the investigator, increases the risks associated with participating in the study such as, a Bazett's corrected QT (QTcB) interval >450 milliseconds (msec).
* Have any lifetime history of a suicide attempt, or have suicidal ideation or, any suicidal behavior within the last month, or who are at significant risk to commit suicide, as judged by the investigator using the Columbia Suicide Severity Rating Scale (C-SSRS).
* Are unsuitable (in the opinion of the investigator or sponsor) for inclusion in the study.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 parts: the open-label, single-dose (SD) period which included 3 cohorts (Cohorts 1 to 3) and the placebo-controlled, multiple-dose (MD) period which included 2 cohorts (Cohorts 4 and 5).
Groups:
- 5 mg LY110140 (SD): Cohort 1: 5-milligram (mg) LY110140 (fluoxetine hydrochloride) capsule orally administered once, in a fasted state, during the SD period.
- 20 mg LY110140 (SD): Cohort 2: 20-mg LY110140 (fluoxetine hydrochloride) capsule orally administered once, in a fasted state, during the SD period.
- 40 mg LY110140 (SD): Cohort 3: 40-mg LY110140 (fluoxetine hydrochloride) dose (two 20-mg LY110140 capsules) orally administered once, in a fasted state, during the SD period.
- Placebo (MD): Participants, in Cohorts 4 and 5, who received a placebo capsule, orally administered once daily for 28 days, during the MD period. On Days 1 and 28 participants were required to fast at least 8 hours prior to dosing and 4 hours postdose.
- 20 mg LY110140 (MD): Participants, in Cohort 4, who received 20-mg LY110140 (fluoxetine hydrochloride) capsule, orally administered once daily for 28 days, during the MD period. On Days 1 and 28, participants were required to fast at least 8 hours prior to dosing and 4 hours postdose.
- 40 mg LY110140 (MD): Participants, in Cohort 5, who received two 20-mg LY110140 (fluoxetine hydrochloride) capsules, orally administered once daily for 28 days, during the MD period. On Days 1 and 28, participants were required to fast at least 8 hours prior to dosing and 4 hours postdose.
Period: Overall Study
Arm/Group | 5 mg LY110140 (SD) | 20 mg LY110140 (SD) | 40 mg LY110140 (SD) | Placebo (MD) | 20 mg LY110140 (MD) | 40 mg LY110140 (MD)
Started | 8 | 8 | 8 | 8 | 12 | 12
Received at Least 1 Dose of Study Drug | 8 | 8 | 8 | 8 | 12 | 12
Completed | 8 | 8 | 8 | 8 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg LY110140 (SD) | 20 mg LY110140 (SD) | 40 mg LY110140 (SD) | Placebo (MD) | 20 mg LY110140 (MD) | 40 mg LY110140 (MD) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 12 | 12 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (4.4) | 25.8 (2.4) | 24.6 (2.4) | 27.1 (4.4) | 25.8 (6.3) | 28.7 (6.2) | 26.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 8 | 12 | 12 | 56
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 8 | 8 | 8 | 8 | 12 | 12 | 56
Region of Enrollment [Number; unit: participants]
  Japan | 8 | 8 | 8 | 8 | 12 | 12 | 56
Cytochrome P450 2D6 (CYP2D6) intermediate and extensive metabolizers [Number; unit: participants] — Based upon a laboratory deoxyribonucleic acid (DNA) screening test, participants were identified as having either the CYP2D6 intermediate metabolizer genotype or the CYP2D6 extensive metabolizer genotype. Intermediate metabolizers were individuals who carry 1 functional (normal or decreased allele) and a null or decreased allele. Extensive metabolizers were individuals with 2 fully active enzyme alleles.
  participants
    CYP2D6 extensive metabolizers | 4 | 4 | 4 | 4 | 6 | 6 | 28
    CYP2D6 intermediate metabolizers | 4 | 4 | 4 | 4 | 6 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug-Related Adverse Events (AEs) or Any Serious AEs During the Single-Dose (SD) Period
Description: A drug-related AE was an AE that occurred postdose or was present predose and became more severe postdose and was considered to be related to study treatment. A summary of AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Day 43
Population: Randomized participants, in Cohorts 1, 2, and 3, who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: participants
Arm/Group | 5 mg LY110140 (SD) | 20 mg LY110140 (SD) | 40 mg LY110140 (SD)
Number analyzed (Participants) | 8 | 8 | 8
participants
  Drug-Related AE | 0 | 0 | 0
  Any Serious AE | 0 | 0 | 0

2. Primary Outcome: Number of Participants With One or More Drug-Related Adverse Events (AEs) or Any Serious AEs During the Multiple-Dose (MD) Period
Description: as for outcome 1
Time Frame: Baseline up to Day 70
Population: Randomized participants, in Cohorts 4 and 5, who received at least 1 dose of study drug or placebo and had at least 1 postdose safety assessment.
Measure: Number; unit: participants
Groups:
- Placebo (MD): Participants, in Cohorts 4 and 5, who received a placebo capsule, orally administered once daily for 28 days, during the MD period. On Days 1 and 28, participants were required to fast at least 8 hours prior to dosing and 4 hours postdose.
Arm/Group | Placebo (MD) | 20 mg LY110140 (MD) | 40 mg LY110140 (MD)
Number analyzed (Participants) | 8 | 12 | 12
participants
  Drug-Related AE | 1 | 0 | 2
  Any Serious AE | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of Single Dose (SD) of LY110140
Description: Study drug was administered as LY110140 (fluoxetine hydrochloride) and its active portion, fluoxetine, was metabolized to norfluoxetine in the body. The Cmax of plasma total fluoxetine and norfluoxetine during the SD period is reported.
Time Frame: Predose up to Day 43
Population: Randomized participants, in Cohorts 1, 2, and 3, who received at least 1 dose of study drug and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 5 mg LY110140 (SD) | 20 mg LY110140 (SD) | 40 mg LY110140 (SD)
Number analyzed (Participants) | 8 | 8 | 8
nanograms per milliliter (ng/mL)
  Fluoxetine | NA (NA) — The fluoxetine concentrations following a single administration of 5 mg LY110140 were below the quantifiable lower limit. | 15.5 (18) | 38.7 (17)
  Norfluoxetine | 2.44 (33) | 13.0 (10) | 22.8 (30)

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Zero to Last Time Point [AUC(0-tlast)] of Single Dose (SD) of LY110140
Description: Study drug was administered as LY110140 (fluoxetine hydrochloride) and its active portion, fluoxetine, was metabolized to norfluoxetine in the body. The AUC(0-tlast) of plasma total fluoxetine and norfluoxetine during the SD period is reported.
Time Frame: Predose up to Day 43
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | 5 mg LY110140 (SD) | 20 mg LY110140 (SD) | 40 mg LY110140 (SD)
Number analyzed (Participants) | 8 | 8 | 8
nanograms*hour per milliliter (ng*hr/mL)
  Fluoxetine | NA (NA) — The fluoxetine concentrations following a single administration of 5 mg LY110140 were below the quantifiable lower limit. | 371 (27) | 1360 (46)
  Norfluoxetine | 195 (74) | 3000 (20) | 5850 (30)

5. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Zero to Infinity [AUC(0-infinity)] of Single Dose (SD) of LY110140
Description: Study drug was administered as LY110140 (fluoxetine hydrochloride) and its active portion, fluoxetine, was metabolized to norfluoxetine in the body. The AUC(0-infinity) of plasma total fluoxetine and norfluoxetine during the SD period is reported.
Time Frame: Predose up to Day 43
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | 5 mg LY110140 (SD) | 20 mg LY110140 (SD) | 40 mg LY110140 (SD)
Number analyzed (Participants) | 8 | 8 | 8
nanograms*hour per milliliter (ng*hr/mL)
  Fluoxetine | NA (NA) — The fluoxetine concentrations following a single administration of 5 mg LY110140 were below the quantifiable lower limit. | 424 (27) | 1430 (46)
  Norfluoxetine | 407 (67) | 3360 (22) | 6360 (32)

6. Secondary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of Multiple Doses (MD) of LY110140
Description: Study drug was administered as LY110140 (fluoxetine hydrochloride) and its active portion, fluoxetine, was metabolized to norfluoxetine in the body. The Cmax of plasma total fluoxetine and norfluoxetine on Day 1 and Day 28 of the MD period is reported.
Time Frame: Days 1 and 28
Population: Randomized participants, in Cohorts 4 and 5, who received at least 1 dose of study drug (excluding placebo) and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 20 mg LY110140 (MD) | 40 mg LY110140 (MD)
Number analyzed (Participants) | 12 | 12
nanograms per milliliter (ng/mL)
  Day 1, Fluoxetine | 16.9 (21) | 39.9 (21)
  Day 28, Fluoxetine | 92.9 (43) | 284 (24)
  Day 1, Norfluoxetine | 10.6 (38) | 18.3 (22)
  Day 28, Norfluoxetine | 136 (28) | 222 (17)

7. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Zero to 24 Hours [AUC(0-24)] of Multiple Doses (MD) of LY110140
Description: Study drug was administered as LY110140 (fluoxetine hydrochloride) and its active portion, fluoxetine, was metabolized to norfluoxetine in the body. The AUC(0-24) of plasma total fluoxetine and norfluoxetine on Day 1 of the MD period is reported.
Time Frame: Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | 20 mg LY110140 (MD) | 40 mg LY110140 (MD)
Number analyzed (Participants) | 12 | 12
nanograms*hour per milliliter (ng*hr/mL)
  Fluoxetine | 228 (29) | 574 (24)
  Norfluoxetine | 199 (41) | 337 (24)

8. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve for Dosing Interval (Tau) at Steady State [AUC(Tau,Steady State)] of Multiple Doses (MD) of LY110140
Description: Study drug was administered as LY110140 (fluoxetine hydrochloride) and its active portion, fluoxetine, was metabolized to norfluoxetine in the body. The AUC(tau,steady state) of plasma total fluoxetine and norfluoxetine during the MD period is reported.
Time Frame: Predose up to Day 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | 20 mg LY110140 (MD) | 40 mg LY110140 (MD)
Number analyzed (Participants) | 12 | 12
nanograms*hour per milliliter (ng*hr/mL)
  Fluoxetine | 1810 (48) | 5910 (25)
  Norfluoxetine | 3010 (29) | 4910 (19)

9. Secondary Outcome: Change From Baseline in Bazett's and Fridericia's Corrected QT (QTcB and QTcF) Intervals
Description: The number of participants with a maximum increase from baseline in 12-lead electrocardiogram (ECG) QTcB and QTcF intervals >30 milliseconds (ms) and >60 ms for the single-dose (SD) and multiple-dose (MD) periods is reported.
Time Frame: Baseline, up to Day 43 (SD period) and Baseline, up to Day 70 (MD period)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 5 mg LY110140 (SD) | 20 mg LY110140 (SD) | 40 mg LY110140 (SD) | Placebo (MD) | 20 mg LY110140 (MD) | 40 mg LY110140 (MD)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 12 | 12
participants
  QTcB >30 ms | 1 | 2 | 2 | 2 | 3 | 6
  QTcF >30 ms | 1 | 0 | 0 | 0 | 1 | 4
  QTcB >60 ms | 0 | 0 | 0 | 0 | 0 | 0
  QTcF >60 ms | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: 5 mg LY110140 (SD) vs 20 mg LY110140 (SD) vs 40 mg LY110140 (SD) vs Placebo (MD) vs 20 mg LY110140 (MD) vs 40 mg LY110140 (MD); Test type: Superiority or Other; Slope = 0.026 — The correlation of time-matched change from baseline QTcF interval (dependent variable) to the time-matched plasma concentration of total fluoxetine and norfluoxetine (covariate) and participant (random effect)

ADVERSE EVENTS:
Groups:
- 20 mg LY110140 (MD): Participants, in Cohort 4, who received 20-mg LY110140 (fluoxetine hydrochloride) capsule, orally administered once daily for 28 days, during the MD period. On Days 1 and 28 participants were required to fast at least 8 hours prior to dosing and 4 hours postdose.
- 40 mg LY110140 (MD): Participants, in Cohort 5, who received two 20-mg LY110140 (fluoxetine hydrochloride) capsules, orally administered once daily for 28 days, during the MD period. On Days 1 and 28 participants were required to fast at least 8 hours prior to dosing and 4 hours postdose.
Arm/Group | 5 mg LY110140 (SD) | 20 mg LY110140 (SD) | 40 mg LY110140 (SD) | Placebo (MD) | 20 mg LY110140 (MD) | 40 mg LY110140 (MD)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/8 | 1/8 | 2/8 | 3/8 | 3/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg LY110140 (SD) (N=8) | 20 mg LY110140 (SD) (N=8) | 40 mg LY110140 (SD) (N=8) | Placebo (MD) (N=8) | 20 mg LY110140 (MD) (N=12) | 40 mg LY110140 (MD) (N=12)
Atrioventricular block first degree (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days